CLINICAL TRIAL: NCT02097147
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group Study Evaluating The Sexual Functioning of Healthy Adults After Receiving Multiple-Dose Regimens of Vilazodone, Paroxetine, or Placebo
Brief Title: Study to Evaluate the Sexual Functioning of Healthy Adults After Receiving Vilazodone, Paroxetine or Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: VLZ-MD-24
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: Viibryd
MeSH Terms: interventions — Vilazodone Hydrochloride; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vilazodone 20 mg (Experimental): Vilazodone 10 mg once daily for 7 days, followed by vilazodone 20 mg once daily for 28 days.
  Interventions: Drug: Vilazodone 20 mg
- Vilazodone 40 mg (Experimental): Vilazodone 10 mg once daily for 7 days, followed by vilazodone 20 mg once daily for 7 days, followed by vilazodone 40 mg once daily for 21 days
  Interventions: Drug: Vilazodone 40 mg
- Paroxetine 20 mg (Active Comparator): Paroxetine 10 mg once daily for 7 days, followed by paroxetine 20 mg for 28 days
  Interventions: Drug: Paroxetine 20 mg
- Placebo (Placebo Comparator): Placebo once daily for 35 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vilazodone 20 mg — Oral administration, once per day.
  Other Names: Viibyrd
  Arms: Vilazodone 20 mg
Drug: Vilazodone 40 mg — Oral administration, once per day.
  Other Names: Viibryd
  Arms: Vilazodone 40 mg
Drug: Paroxetine 20 mg — Oral administration, once per day.
  Other Names: Paxil
  Arms: Paroxetine 20 mg
Drug: Placebo — Oral administration, once per day.
  Arms: Placebo

SUMMARY:
To compare the effects of vilazodone, paroxetine and placebo on sexual function in sexually active healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, aged 18 through 45 years, inclusive
* Currently sexually active
* If female, non pregnant and agree to use acceptable for of contraception during
* If male, be sterile or have partner use contraception.

Exclusion Criteria:

* Have sexual dysfunction
* Have history of diagnosis or treatment of any disorder related to sexual functioning.
* Clinically significant disease state, in the opinion of the examining physician, in any body system
* History of alcohol or other substance abuse or dependence within the previous 5 years

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Changes in Sexual Functioning Questionnaire (CSFQ) total score | From Baseline to Day 35
  The CSFQ is a subject-rated scale designed to measure changes in sexual function and is a structured, self-report, 14-item questionnaire, that measures sexual functioning as a total score (all 14 items), and on the subscales of pleasure, desire/frequency, desire/interest, arousal, and orgasm, rated on a 5 point scale, with each item rated from 1 to 5, and a total score range of 14 to 70. Lower scores are associated with worsened sexual functioning.

SECONDARY OUTCOMES:
Proportion of subjects meeting criteria for sexual dysfunction. | 5 Weeks
  Proportion of subjects meeting criteria for sexual dysfunction (ie, CSFQ <=47 for males and <=41 for females) at any 2 consecutive visits during the double-blind treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Maju Mathews, MD, Study Director — Forest Laboratories
Locations (4):
- United States (4):
  - Forest Investigative Site 001, Miami, Florida
  - Forest Investigative Site 002, Overland Park, Kansas
  - Forest Investigative Site 003, Saint Paul, Minnesota
  - Forest Investigative Site 004, Charlottesville, Virginia